CLINICAL TRIAL: NCT00122941
Title: Effect of Multiple Micronutrient Supplementation on Growth, Morbidity, and Mortality of HIV Infected Children in Uganda: a Randomised Double Blind Placebo-Controlled Trial
Brief Title: Effect of Multiple Micronutrient Supplementation on Growth, Morbidity, and Mortality of HIV Infected Children in Uganda
Acronym: MMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: The Norwegian Programme for Development, Research and Higher Education (Other)
Responsible Party: James K Tumwine, Makerere University Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2002/HD11/2078/MMS; MV910
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: multiple; micronutrients; supplementation; HIV; children; randomised; trial; mortality; morbidity; growth; Uganda
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: multiple micronutrients

SUMMARY:
Micronutrient deficiencies are common in HIV infected children and are aggravated by poor nutrition, especially in poor resource countries such as Uganda. It appears that micronutrient deficiencies contribute to immune dysfunction, increased morbidity and HIV disease progression. Hitherto, there has been no randomised controlled trial to assess the effect of multiple micronutrient supplementation on morbidity and mortality in HIV infected children in Africa. Therefore, the investigators shall carry out a randomised controlled trial to determine the effect of multiple micronutrient supplementation on morbidity, weight gain and mortality among HIV infected children aged 1 to 5 years in Uganda.

Hypothesis: Daily administration of twice the recommended dietary allowance (2RDA) of multiple micronutrients to HIV infected children aged one to five years, for 6 months, will reduce all cause mortality from 24% to 14.4% in one year and result in a weight gain difference of 150 grams.

DETAILED DESCRIPTION:
Micronutrient deficiencies are common in HIV infected children and are aggravated by poor nutrition, especially in poor resource countries such as Uganda. It appears that micronutrient deficiencies contribute to immune dysfunction, increased morbidity and HIV disease progression. Hitherto, there has been no randomised controlled trial to assess the effect of multiple micronutrient supplementation on morbidity and mortality in HIV infected children in Africa. Therefore, the investigators shall carry out a randomised controlled trial to determine the effect of multiple micronutrient supplementation on morbidity, weight gain and mortality among HIV infected children aged 1 to 5 years in Uganda.

Hypothesis: Daily administration of twice the recommended dietary allowance (2RDA) of multiple micronutrients to HIV infected children aged one to five years, for 6 months, will reduce all cause mortality from 24% to 14.4% in one year and result in a weight gain difference of 150 grams.

A sample size of 373 was calculated assuming that the mortality risk in one year in HIV infected children is 24% (Barhane et al) and that this risk will be reduced to 14.4% in the intervention group (40% effect size) with 90% power and 95% confidence.

Assuming a 10% attrition rate (38 study participants), the final sample size in each group is 411.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to 5 years
* HIV infection (previously confirmed by 2 ELISAs for children > 18 months; DNA PCR for those < 18 months)
* Informed consent from the parent/caretaker
* Ability to return for follow-up (lives within a radius of 15 km from hospital and unlikely to change residence during the course of the study)

Exclusion Criteria:

* Children already enrolled in other studies
* Children with severe abnormalities which are likely to impair oral intake (for example, severe cerebral palsy)
* Severely ill children requiring urgent admission and resuscitation

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 860 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of children dying during the study period
Average weight gain in each of the treatment groups

SECONDARY OUTCOMES:
Blood micronutrient levels
Incidence/prevalence of diarrhoea
HIV disease progression (CD4 count and clinical staging)
Prevalence of C. parvum and E. bieneusi
Adverse events related to supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Grace Ndeezi, MMed, Principal Investigator — Makerere University, Medical School, Department of Paediatrics and Child Health
Locations (2):
- Centre for International Health University of Bergen, Bergen, Bergen, Norway
- Department of Paediatrics and Child Health, Mulago Hospital, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Jiamton S, Pepin J, Suttent R, Filteau S, Mahakkanukrauh B, Hanshaoworakul W, Chaisilwattana P, Suthipinittharm P, Shetty P, Jaffar S. A randomized trial of the impact of multiple micronutrient supplementation on mortality among HIV-infected individuals living in Bangkok. AIDS. 2003 Nov 21;17(17):2461-9. doi: 10.1097/00002030-200311210-00008. PMID 14600517
- [Background] Kelly P, Musonda R, Kafwembe E, Kaetano L, Keane E, Farthing M. Micronutrient supplementation in the AIDS diarrhoea-wasting syndrome in Zambia: a randomized controlled trial. AIDS. 1999 Mar 11;13(4):495-500. doi: 10.1097/00002030-199903110-00008. PMID 10197378
- [Background] Bhutta ZA, Black RE, Brown KH, Gardner JM, Gore S, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Prevention of diarrhea and pneumonia by zinc supplementation in children in developing countries: pooled analysis of randomized controlled trials. Zinc Investigators' Collaborative Group. J Pediatr. 1999 Dec;135(6):689-97. doi: 10.1016/s0022-3476(99)70086-7. PMID 10586170
- [Background] Campa A, Shor-Posner G, Indacochea F, Zhang G, Lai H, Asthana D, Scott GB, Baum MK. Mortality risk in selenium-deficient HIV-positive children. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Apr 15;20(5):508-13. doi: 10.1097/00042560-199904150-00015. PMID 10225235
- [Background] Tang AM, Graham NM, Semba RD, Saah AJ. Association between serum vitamin A and E levels and HIV-1 disease progression. AIDS. 1997 Apr;11(5):613-20. doi: 10.1097/00002030-199705000-00009. PMID 9108943
- [Background] Allard JP, Aghdassi E, Chau J, Tam C, Kovacs CM, Salit IE, Walmsley SL. Effects of vitamin E and C supplementation on oxidative stress and viral load in HIV-infected subjects. AIDS. 1998 Sep 10;12(13):1653-9. doi: 10.1097/00002030-199813000-00013. PMID 9764785
- [Background] Fawzi W, Msamanga G, Spiegelman D, Hunter DJ. Studies of vitamins and minerals and HIV transmission and disease progression. J Nutr. 2005 Apr;135(4):938-44. doi: 10.1093/jn/135.4.938. PMID 15795466
- [Derived] Ndeezi G, Tumwine JK, Ndugwa CM, Bolann BJ, Tylleskar T. Multiple micronutrient supplementation improves vitamin B(1)(2) and folate concentrations of HIV infected children in Uganda: a randomized controlled trial. Nutr J. 2011 May 21;10:56. doi: 10.1186/1475-2891-10-56. PMID 21600005
- [Derived] Ndeezi G, Tumwine JK, Bolann BJ, Ndugwa CM, Tylleskar T. Zinc status in HIV infected Ugandan children aged 1-5 years: a cross sectional baseline survey. BMC Pediatr. 2010 Sep 21;10:68. doi: 10.1186/1471-2431-10-68. PMID 20858275
- [Derived] Ndeezi G, Tylleskar T, Ndugwa CM, Tumwine JK. Effect of multiple micronutrient supplementation on survival of HIV-infected children in Uganda: a randomized, controlled trial. J Int AIDS Soc. 2010 Jun 3;13:18. doi: 10.1186/1758-2652-13-18. PMID 20525230